CLINICAL TRIAL: NCT03811730
Title: The Diagnosis and Treatment System of Transesophageal Echocardiography in ICU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kang Yan (Other)
Responsible Party: Sponsor-Investigator, Kang Yan, Director, West China Hospital
Organization: West China Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: TEE
Record Dates: First submitted 2019-01-10; First posted 2019-01-22 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: Critically Ill
Keywords: transesophageal echocardiography; intensive care unit
MeSH Terms: conditions — Critical Illness | interventions — Echocardiography, Transesophageal; Echocardiography

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TEE group (Experimental): Eligible patients would be conducted TEE examination by researcher A,The examination results are judged by A and provided to the physician of this patient,
  Interventions: Diagnostic Test: Transesophageal echocardiography
- TTE group (Active Comparator): Eligible patients would be conducted TTE examination by researcher B,The examination results are judged by B and provided to the physician of this patient,
  Interventions: Diagnostic Test: Transesophageal echocardiography

INTERVENTIONS:
Diagnostic Test: Transesophageal echocardiography — Eligible patients would be conducted both Transesophageal echocardiography and Transthoracic echocardiography to offer independent results
  Other Names: Transthoracic echocardiography

SUMMARY:
Transesophageal ultrasound offers imaging through the esophagus on the surface of the heart, with good image quality and unique advantages. However, no studies to date have examined its effect in critically ill patients in China.Therefore, the investigators aimed to compare the efficacy and safety of TEE with TTE. the investigators will conducte a Multi-center, prospective observational control study enrolling critically ill adult patients in several ICU in China .

DETAILED DESCRIPTION:
Patients in ICU were assessed for the need for TEE by trained researcher. Eligible patients would be conducted tee examination by researcher A, TTE by the researcher B ,at the same time, researcher C records the basic condition and clinical data of patientsand carried out micro-enlargement test.The examination results are judged by A and B respectively and provided to the physician of this patient, and A return visit to the physician wold be conducted by researcher D to evaluate the acceptance of TTE and TEE results and judge the clinical effects. The primary outcome is the clinical effects.

ELIGIBILITY:
Inclusion Criteria:

1. The quality of Transthoracic echocardiography is poor ( >3 sections cannot be obtained or the inner membrane is not clear)
2. The diagnosis of the etiology by Transthoracic ultrasonography is still unclear
3. The results of Transthoracic ultrasonography are inconsistent with clinical judgment or cannot explain the existing signs.
4. No obvious improvement or even aggravation after thoracic examination and corresponding treatment
5. Special conditions or clinical scenarios
6. Other clinicians think a TEE check is required.

Exclusion Criteria:

1. There is a tee test taboo and clinicians evaluate the risk over benefit
2. Did not sign an informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Conclusion of the adoption | 48 hours after completion of the examination
  Researcher C conducted a questionnaire survey on attending physician to evaluate the effect

SECONDARY OUTCOMES:
adverse events | completion of the examination
  Adverse events associated with the examination，eg.1.Anesthetic allergy;2.Nausea, vomiting, choking cough or aspiration;3.Laryngeal edema and even asphyxiation;4.Severe arrhythmia;5.Esophageal perforation, bleeding, or local hematoma;6.Other accidental deaths, such as acute myocardial infarction, shock, haemorrhage and possibly even death;7.Other unpredictable contingencies or complications

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Department of Critical Care Medicine, Peking Union Medical College Hospital, Peking Union Medical College & Chinese Academy of Medical Sciences, Beijing
  - Xiangya Hospital Central South University, Changsha
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning
  - The First Hospital of China Medical University, Shengyang
  - Zhongnan Hospital of Wuhan University, Wuhan